CLINICAL TRIAL: NCT01535196
Title: Effects of 25-OH-D3 Vitamin Substitution in Congestive Heart Failure. Controlled, Randomized, Double Blind Trial
Brief Title: Vitamine D Treatment in Chronic Heart Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: financial reasons / insufficient enrollment activity
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Istvan Takacs, Principal investigator, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-heart
Record Dates: First submitted 2012-01-09; First posted 2012-02-17 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Chronic Heart Failure; Vitamin D Adverse Reaction
Keywords: vitamin D; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25-OH-D3 vitamin (Experimental): 180 000 IU 25-OH-D3 vitamin oil per os, per month in the 0, 1, 2, 3, and 6 month at the visit. The patient take the drug under medical control
  Interventions: Drug: Vigantol oil and MCT oil
- MCT oil (Placebo Comparator): 9 ml MCT oil as placebo in the 0,1,2,3,6 month at the visit, under medical contol
  Interventions: Drug: Vigantol oil and MCT oil

INTERVENTIONS:
Drug: Vigantol oil and MCT oil — Vigantol oil, 9 ml, 180 000 IU at the 0,1,2,3,6 month (5 times in the study) MCT oil as placebo, 9 ml, 0,1,2,3,6 month (5 times in the study)
  Other Names: no other name

SUMMARY:
The investigators hypothesized that in vitamin D deficiency the 25-OH-D3 vitamin substitution improve the heart function in chronic heart failure.

Type of study: Controlled, randomized, double blind, placebo control

Number of patient: 300; 150 treated and 150 placebo controlled

Type of drug: 180 000 IU 25-OH-D3 vitamin oil (Vigantol) per month in the 0,1,2,3,6, month

Duration of study:1+1 year

Primary end points:

Survival rate, Ejection fraction by ultrasound, Brain natriuretic peptid,

Secondary end points:

Safety of D-vitamin supplementation, well being score, blood pressure, BMI Walking distant in 6 minutes

Visits:

Screening, Randomization, 1month, 2 month, 3 month, 6 month, 12 month, 24 month,

ELIGIBILITY:
Inclusion Criteria:

* NYHA II-IV
* vitamin D level between 10-30 ng/ml
* ejection fraction by ultrasound < 40 %

Exclusion Criteria:

* blood calcium > 2,6 mmol/l
* urinary calcium > 0,1 mmol/body weight kg/die
* blood phosphorus > 1,45 mmol/l
* nephrolithiasis in the history
* GFR < 30 ml/min
* vitamin D injection in the last 6 month
* actual 1,25-OH2-D3 vitamin treatment
* Myocardial infarction or serious coronaria stenosis in the anamnesis uncontrolled atrial fibrillation
* serious valve disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Survival rate | 2 years

SECONDARY OUTCOMES:
D-vitamin supplementation safety | 1 year
ejection fraction by ultrasound | 2 years
serum brain natriuretic peptid level | 2 years
walking test in 6 minutes | 2 years
well-being score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Takacs, PhD, Principal Investigator — Semmelweis University
Locations (2):
- Hungary (2):
  - Semmelweis University Ist Department of Medicine, Budapest
  - Semmelweis University Cardiovascular Center, Budapest